CLINICAL TRIAL: NCT04852926
Title: Study of the Sexual Health of Patients Treated for Non-metastatic Breast Cancer and Followed up in the Observatory of Fertility at Jeanne de Flandre Hospital : a Prospective Monocentric Cohort With Repeated Anonymous Self-administered Questionnaires.
Brief Title: Study of the Sexual Health of Patients Treated for Breast Cancer and Followed up in the Observatory of Fertility at Jeanne de Flandre Hospital.
Acronym: ENVIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_61; 2020-A00541-40 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Carcinoma; Breast Tumor
Keywords: Breast cancer; Fertility preservation Quality of life Sexual health Marital satisfaction; Quality of life; Sexual health; Marital satisfaction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A prospective cohort of patients: Female patients treated for non-metastatic breast cancer and followed up in the Observatory of fertility at Jeanne de Flandre Hospital
  Interventions: Other: Self-administered questionnaires

INTERVENTIONS:
Other: Self-administered questionnaires — 6 self-administered questionnaires (EORTC-QLQ-C30, RSE, BIS, HAD, FSFI, DAS-4) completed by the patients at every usual follow-up consultation.
  1 (FSFI) or 2 (MSHQ, PEP) self-administered questionnaires completed by the partner (respectively female or male) between every usual follow-up consultation.
  Follow-up usual consultations :
  * T0 (at inclusion) : before disease + since diagnosis
  * C4 (chemotherapy course n°4)
  * C6 (chemotherapy course n°6)
  * M3 (3 months after chemotherapy)
  * M6 (6 months after chemotherapy)
  * A1 (1 year after chemotherapy)
  * A2 (2 years after chemotherapy)

SUMMARY:
Study of sexual health by repeated anonymous self-administered questionnaires in patients treated for non-metastatic breast cancer and referred to Jeanne de Flandre hospital for possible preservation of their fertility. Sexual health is affected by treatments and improves after the treatments. Sexual health is influenced by multiple factors : oncology treatments received, self-esteem, body image, anxiety, depression, professional activity

ELIGIBILITY:
Inclusion Criteria:

* Female from 18 years
* In a relationship with a man or a woman
* Developing invasive carcinoma of breast cancer
* Planned medical therapy project by chemotherapy
* Followed up in the Observatory of fertility
* Patient who gave written consent to participate in the study
* Insured Social Patient
* Patient willing to follow all study procedures and duration

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients treated for non-metastatic breast cancer and followed up in the Observatory of fertility at Jeanne de Flandre Hospital.
Study Population: * Refusal of oncologic treatments
  * Other cancer than breast cancer
  * Metastatic breast cancer
  * Unable to receive informed information, unable to participate in the entire study, lack of social security coverage, refusal to sign consent
  * Person under protection
  * Minor
  * Persons deprived of liberty
  * Persons unable to consent
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
variation of score FSFI (female sexual function index) | At 1 year after the start of chemotherapy
  The FSFI score assesses female sexual functioning over the past four weeks. It is a self-evaluation by questionnaire. It consists of 19 questions with 5 or 6 possible answers per question, scored respectively from 1 to 5 and from 0 To evaluate, in women with non-metallic breast cancer followed in the Fertility Observatory at the Jeanne de Flandre Hospital, 1-year sexual health progression from chemotherapy initiation to sexual health assessment prior to cancer diagnosis announcement.

SECONDARY OUTCOMES:
evolution of quality of life and psychometric factors at 1 year from the start of chemotherapy compared to the evaluation of these factors before the cancer diagnosis is announced. | At inclusion, at 1 year and 2 years after chemotherapy
association between psychometric factors assessed prior to cancer diagnosis and sexual health progression at 1 year of chemotherapy initiation | At inclusion, at 1 year and 2 years after chemotherapy
correlation between quality of life and psychometric factors and the assessment of sexual health of patients measured at all times. | At inclusion, at 1 year and 2 years after chemotherapy
describe partners' sexual health by MSHQ (man)/FSFI (woman) during follow-up | At inclusion, at chemotherapy course n°4, at chemotherapy course n°6, at 3 months and at 6 months after chemotherapy, at 1 year and 2 years after chemotherapy,
  MSHQ (Male Sexual Health Questionnaire) consists of 25 questions. It is a self-evaluation by the partner. A total score out of 125 is calculated. A high score corresponds to a good quality of male sexual life.
describe partners' sexual health by PEP (man)/FSFI (woman) during follow-up | At inclusion, at chemotherapy course n°4, at chemotherapy course n°6, at 3 months and at 6 months after chemotherapy, at 1 year and 2 years after chemotherapy,
  The PEP (Premature ejaculation profile) score explores premature ejaculation by self-questionnaire. It consists of 4 questions scored from 1 to 5. A high score corresponds to good male sexual health. A low score indicates premature ejaculation with repercussions on male sexual health.
testimony of patients expressing their experience of follow-up in the Fertility Observatory | At inclusion, at chemotherapy course n°4, at chemotherapy course n°6, at 3 months and at 6 months after chemotherapy, at 1 year and 2 years after chemotherapy,

CONTACTS AND LOCATIONS:
Overall Officials: Carine Martin, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France